CLINICAL TRIAL: NCT01347879
Title: PCTA206/11 A Double Blinded, Prospective, Randomized, Vehicle Controlled Multi Center Study of Photodynamic Therapy With Visonac® Cream in Patients With Acne Vulgaris.
Brief Title: A Double Blinded, Prospective, Randomized, Vehicle Controlled Multi-center Study of Photodynamic Therapy With Visonac® Cream in Patients With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Photocure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCTA206/11
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-12

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; PDT
MeSH Terms: conditions — Acne Vulgaris | interventions — Red Light; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visonac cream with PDT (Experimental): active treatment with light dose of 37 Joule/cm2
  Interventions: Drug: Visonac PDT
- Vehicle cream with PDT (Placebo Comparator): Placebo treatment, Light dose 37 Joule/cm2
  Interventions: Drug: Vehicle cream with PDT

INTERVENTIONS:
Drug: Visonac PDT — cream application prior to illumination with red light
  Other Names: red light
  Arms: Visonac cream with PDT
Drug: Vehicle cream with PDT — placebo/vehicle cream application prior to illumination with red light
  Other Names: red light
  Arms: Vehicle cream with PDT

SUMMARY:
This study is intended to evaluate the efficacy and safety of Visonac Photodynamic Therapy (PDT) in patients with severe acne, score 4 on global IGA scale. The null hypothesis is that Visonac PDT is equal to vehicle PDT against the alternative hypothesis that Visonac PDT is different compared to vehicle PDT at week 12.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients, from 12-35 years of age with severe facial acne vulgaris (IGA score 4 on IGA scale)
* Signed and verified informed consent form and photo consent form. For subjects under age of 18, an assent form in conjunction with an informed consent form, signed and verified by parent/guardian.
* Female patients who are surgically sterile, pre-menstrual, postmenopausal, abstinent, or willing to use an adequate means of contraception including birth control pills, or barrier methods and spermicide for at least 14 days prior to T1. Patients using birth control pills must have used the same product and dose for at least 3 months and must agree to stay with the same product and dose for an additional 3 months.
* Fitzpatrick skin type I through VI,
* Patients with 25 to 75 inflammatory lesions (papules, pustules, and nodules) on the face.
* Patients with 20 to 100 non-inflammatory lesions (open and closed comedones) on the face.

Exclusion Criteria:

* Patients with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.)
* Patients with more than 3 nodules on the face.
* Patient is the investigator or any sub investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
* Patients unlikely to comply with the protocol, e.g. mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the clinical study, uncooperative attitude or unlikelihood of completing the study (e.g. drug or alcohol abuse).
* Female patients with childbearing potential (i.e. ovulation, pre-menopausal, not surgically sterilized) and sexually active, not willing to use a medically accepted contraceptive regimen (as described under inclusion criteria) while on treatment.
* Pregnancy.
* Nursing.
* Participation in other clinical studies either currently or within the last 30 days.
* Patients with porphyria.
* Patients with cutaneous photosensitivity.
* Known allergy to MAL, to a similar PDT compound, or to excipients of the cream
* Patients using testosterone, any other systemic hormonal treatment or hormonal contraceptives solely for control of acne.
* Patients who have received topical treatments for their facial acne within the last 14 days (e.g steroids, retinoids, glycolic acid, benzoyl peroxide, anti inflammatory agents, antibiotics). Medicated cleansers may be used during the washout period and stopped before the treatment.
* Patients who have received oral antibiotics for treatment of their acne within the last month.
* Patients who have received oral isotretinoin within the last 6 months.
* Patient who have received facial procedures like dermabrasion, chemical or laser peels within the last 1 month.
* Patients using testosterone, any systemic hormonal treatment for other reasons than acne treatment and has not been on the same product and dose for at least 3 months
* Patients with moderate, severe or very severe facial acne scarring according to scarring scale described in section 10.4.3.
* Patients with a beard that might interfere with study assessments.
* Patients with melanoma or dysplastic nevi in the treatment area.
* Exposure to ultraviolet radiation (UVB phototherapy, sun tanning salons) within the last 30 days
* Exposure to PDT within 12 weeks before T1.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2011-05; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Pariser, MD, Principal Investigator — Virginia Clinical Research, Inc.
Locations (15):
- United States (15):
  - Dermatology Specialists Inc, Oceanside, California
  - Rady Children's Hospital, San Diego, California
  - North Florida Dermatology Associates, Jacksonville, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Dermatology Institute, DuPage Medical Group, Naperville, Illinois
  - Deaconess Clinic Inc, Evansville, Indiana
  - ActivMed Practices & Research Inc, Haverhill, Massachusetts
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Clinical Partners LLC, Johnston, Rhode Island
  - DermResearch Inc, Austin, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dermatology clinics in the US.
Groups:
- Vehicle Cream With PDT: Placebo treatment, Light dose 37 J/cm2
  Visonac PDT : cream application prior to illumination with red light
- Visonac Cream With PDT: active treatment with light dose of 37 J/cm2
  Visonac photodynamic therapy (PDT): cream application prior to illumination with red light
Period: Overall Study
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Started | 53 | 100
Completed | 46 | 83
Not Completed | 7 | 17
Not completed — Adverse Event | 0 | 12
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Visonac Cream With PDT: active treatment with light dose of 37J/cm2
  Visonac PDT : cream application prior to illumination with red light
- Total: Total of all reporting groups
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT | Total
Number analyzed (Participants) | 53 | 100 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 59 | 94
  Between 18 and 65 years | 18 | 41 | 59
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.6 (5.8) | 18.6 (5.5) | 18.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 44 | 66
  Male | 31 | 56 | 87
Region of Enrollment [Number; unit: participants]
  United States | 53 | 100 | 153
Skin type [Number; unit: participants] — Fitzpatrick skin type. The Fitzpatrick Scale:
  Type I (scores 0-7) Light, pale white. Always burns, never tans
  Type II (scores 8-16) White; fair. Usually burns, tans with difficulty
  Type III (scores 17-24) Medium, white to olive. Sometimes mild burn, gradually tans to olive.
  Type IV (scores 25-30) Olive, moderate brown. Rarely burns, tans with ease to a moderate brown.
  Type V (scores over 30) Brown, dark brown. Very rarely burns, tans very easily
  Type VI Black, very dark brown to black. Never burns, tans very easily, deeply pigmented.
  participants
    Skin type I | 0 | 1 | 1
    Skin type II | 24 | 34 | 58
    Skin type III | 15 | 38 | 53
    Skin type IV | 7 | 15 | 22
    Skin type V | 6 | 8 | 14
    Skin type VI | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Facial Inflammatory Lesion Count (Nodules, Papules, and Pustules).
Time Frame: From baseline to 12 weeks after first treatment
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
lesion count | -7.8 (21.4) | -15.6 (16.4)
Statistical Analysis 1: Comparison: Vehicle Cream With PDT vs Visonac Cream With PDT; Test type: Superiority or Other; p = 0.006, ANCOVA; Lesion count at baseline and center as covariates; Difference in least square means = -7.35, 95% CI 2-sided [-12.5 to -2.2]

2. Secondary Outcome: Absolute Change From Baseline in Facial Non-inflammatory Lesion Count (Open and Closed Comedones)
Time Frame: From baseline to 12 weeks after the first treatment
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
lesion count | -10.7 (22.1) | -11.8 (19.0)
Statistical Analysis 1: Comparison: Vehicle Cream With PDT vs Visonac Cream With PDT; Test type: Superiority or Other; p = 0.8527, ANCOVA; Lesion count at baseline and center as covariates; Difference in least square means = -0.6, 95% CI 2-sided [-6.6 to 5.5]

3. Secondary Outcome: Percent Change From Baseline in Facial Inflammatory (Nodules, Papules, and Pustules)Lesion Counts.
Time Frame: From baseline to 12 weeks after the first treatment
Measure: Median (Full Range); unit: percent change
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
percent change | -26.6 [-100 to 176] | -43.8 [-100 to 84]
Statistical Analysis 1: Comparison: Vehicle Cream With PDT vs Visonac Cream With PDT; Test type: Superiority or Other; p = 0.0032, ANCOVA; Lesion count at baseline and center as covariates; Difference in least square means = -20.0, 95% CI 2-sided [-33.2 to -6.8]

4. Secondary Outcome: Proportion of Patients With Success According to IGA Scale Based on the Facial Assessment.
Description: One Investigator Global Assessment (IGA) scale was used including inflammatory and non-inflammatory lesions. The investigator qualitatively graded the overall acne severity on a scale from 0 to 4, with 4 being the most severe. Success was defined as an improvement of at least 2 grades from the baseline score.
Time Frame: From baseline to 12 weeks after first treatment
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
participants | 14 | 44
Statistical Analysis 1: Comparison: Vehicle Cream With PDT vs Visonac Cream With PDT; Test type: Superiority or Other; p = 0.0125, Regression, Logistic

5. Secondary Outcome: Pain During Illumination.
Description: Pain during illumination was assessed by patient using a Visual Analogue Scale (VAS) from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable.
Time Frame: Immediately after first treatment
Measure: Mean (Full Range); unit: VAS score in cm
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
VAS score in cm | 0.52 [0.0 to 3.6] | 3.38 [0.0 to 8.8]

6. Secondary Outcome: Number of Patients With Adverse Events.
Time Frame: From administration of investigational medicinal product (IMP) until 12 weeks after first IMP administration
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
participants | 14 | 48

7. Secondary Outcome: Erythema Score of Mild and Moderate
Description: Clinical assessment using a 4 point scale; none, mild, moderate, severe
Time Frame: Immediately after first treatment
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
participants | 37 | 86

8. Secondary Outcome: Clear and Almost Clear Scarring According to Scarring Score
Description: Clinical assessment using a 6 point scale; Clear, Almost clear, Mild, Moderate, Severe and Very severe
Time Frame: at week 12 after first treatment
Population: 100 patients were included and 83 patients completed the study in the Visonac treatment arm. However, a few patients came back for the week 12 visit only, and have data for scarring. The total number of patients with scarring data at 12 weeks in this group is 91.
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 46 | 91
participants | 25 | 53

9. Secondary Outcome: Percent Change From Baseline in Facial Non-inflammatory Lesion Count (Open and Closed Comedones)
Time Frame: From baseline to 12 weeks after first treatment
Measure: Median (Full Range); unit: percent change
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
percent change | -37.0 [-100 to 196] | -31.0 [-100 to 100]
Statistical Analysis 1: Comparison: Vehicle Cream With PDT vs Visonac Cream With PDT; Test type: Superiority or Other; p = 0.7161, ANCOVA; Lesion count at baseline and center as covariate; Difference in least square means = -2.56, 95% CI 2-sided [-16.5 to 11.3]

10. Secondary Outcome: Erythema Score of Severe
Description: Clinical assessment using a 4 point scale; none, mild, moderate, severe
Time Frame: Immediately after first treatment
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 100
participants | 0 | 3

11. Secondary Outcome: Erythema Score of Mild and Moderate
Description: Clinical assessment using a 4 point scale; none, mild, moderate, severe
Time Frame: 2 days after first treatment
Population: Of the 100 patients who were included in the Visonac treatment arm, 5 dropped out prior to the day 2 erythema assessment. The number of patients with erythema data at this assessment point is 95.
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 95
participants | 26 | 65

12. Secondary Outcome: Erythema Score of Severe
Description: Clinical assessment using a 4 point scale; none, mild, moderate, severe
Time Frame: 2 days after first treatment
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 53 | 95
participants | 0 | 0

13. Secondary Outcome: Mild and Moderate Scarring According to Scarring Score
Description: Clinical assessment using a 6 point scale; Clear, Almost clear, Mild, Moderate, Severe and Very severe
Time Frame: at week 12 after first treatment
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 46 | 91
participants | 21 | 38

14. Secondary Outcome: Severe and Very Severe Scarring According to Scarring Score
Description: Clinical assessment using a 6 point scale; Clear, Almost clear, Mild, Moderate, Severe and Very severe
Time Frame: at week 12 after first treatment
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Number analyzed (Participants) | 46 | 91
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Vehicle Cream With PDT | Visonac Cream With PDT
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/100
Other Adverse Events (participants affected / at risk) | 14/53 | 48/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Cream With PDT (N=53) | Visonac Cream With PDT (N=100)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 17
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 8
Erythema (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Scab (Skin and subcutaneous tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Conjunctivitis bacterial (Eye disorders) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth abscess (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (General disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less